CLINICAL TRIAL: NCT02709317
Title: Preventing Risky Drinking in Veterans Treated With Prescription Opioids
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Collaborators: United States Department of Defense (U.S. Federal Agency); Corporal Michael J. Crescenz VA Medical Center (U.S. Federal Agency); Medical University of South Carolina (Other); VA Pittsburgh Healthcare System (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 818671
Record Dates: First submitted 2016-01-28; First posted 2016-03-16 (Estimated); Results first posted 2022-03-02 (Actual); Last update posted 2022-03-02 (Actual); Status verified 2021-12

CONDITIONS: Pain; Opiates; Alcohol Drinking
MeSH Terms: conditions — Pain; Alcohol Drinking | interventions — Crisis Intervention

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Standard Care (Active Comparator): In this arm, veterans receive the care that they would receive had they not enrolled in the research. No one will receive less than standard care.
  Interventions: Behavioral: Brief Intervention
- Prevention Intervention (Experimental): An adaptive monitoring intervention, delivered through text messages and brief telephone calls, that can provide extended prevention services for veterans engaging in risky alcohol use. After a veteran receives a BI for risky drinking, we will monitor alcohol use for 4 weeks. Veterans who reduce alcohol use to safe levels will be placed in a monitoring track, which consists of tailored text messages and brief monthly telephone contacts. Conversely, veterans who continue to use alcohol at hazardous levels will be placed in a track that provides tailored text messages and more frequent telephone calls. These calls provide further prevention/intervention services to help the veteran reduce alcohol use. These services address motivational issues and identify more effective ways to cope with stress and other factors that trigger unsafe alcohol use. Information on the veteran's progress is used to guide the content of subsequent text messages and prevention interventions.
  Interventions: Behavioral: Prevention Intervention; Behavioral: Brief Intervention

INTERVENTIONS:
Behavioral: Prevention Intervention
  Arms: Prevention Intervention
Behavioral: Brief Intervention

SUMMARY:
Veterans who are taking prescription opioids for chronic pain and are engaging in risky drinking are at heightened risk for drug interactions, including overdose and other negative effects, particularly if they are also using benzodiazepines. The investigators propose to test a prevention intervention, designed to reduce rates of risky drinking in veterans receiving prescription opioids to treat their chronic pain. This adaptive, patient-centered intervention provides clinical assessment, brief intervention, monitoring, and extended prevention services delivered through a combination of clinical visits, telephone calls, and text messages. The investigators propose to conduct a study in which veterans (N=300) who are on daily doses of prescription opioids will be randomized to receive 12 months of an adaptive prevention intervention (PI) or to standard care (SC), which consists of a Brief Intervention (BI) with 2 follow-up contacts. Potential participants will be veterans at the Philadelphia VA, and surrounding areas, or the Pittsburgh VA who, based on pharmacy records, are using opioids daily to treat chronic pain. An initial evaluation will identify individuals who also engage in risky alcohol use based on NIAAA-recommended guidelines and meet other inclusion criteria to be enrolled in the study. The evaluation will also identify the use of other medications (e.g., benzodiazepines) that could interact negatively with opioid use. For veterans randomized to the PI condition, a BI is first provided to reduce alcohol to non-hazardous levels and the effects are monitored for one month. Veterans who reduce alcohol use to non-hazardous levels during this one-month period continue in a monitoring track, consisting of tailored text messages and brief monthly telephone contacts. Veterans who continue to drink at risky levels are instead placed in a track that provides tailored text messages and more frequent telephone calls. In addition to monitoring, these calls provide further prevention/BI services to help the veteran reduce alcohol use to non-hazardous levels. Key components of these services are motivational enhancement and development of more effective ways to cope with stress and other triggers for risky alcohol use. All participants will be followed up at 3, 6, 9, 12 and 18 months after baseline. The primary outcome at each follow-up point will be a dichotomous measure of any risky drinking since the prior follow-up (yes/no). Secondary outcomes will include self-reported frequency of heavy drinking, biological measures of alcohol use, other drug use as determined by urine toxicology tests, opioid overdoses, and ratings of depression and pain. Repeated measures analyses will compare the PI and SC conditions on primary and secondary outcomes assessed across an 18-month follow-up. Analyses will also test hypothesized moderation and mediation effects.

ELIGIBILITY:
Inclusion Criteria:

* currently be receiving daily treatment with a prescription opioid for chronic pain;
* be 18 years or older;
* have a cell phone capable of receiving text messages;
* and be willing to be in a study where they might receive text messages.

Exclusion Criteria:

* meet DSM-V criteria for a moderate to severe alcohol or drug disorder (with the exception of nicotine abuse/dependence);
* have a current psychotic disorder severe enough to require inpatient treatment;
* are participating in substance abuse treatment at the VA or elsewhere (with exception of screening and brief intervention at the VA).

Ages: 18 Years to 88 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 108 (Actual)
Dates: Start 2014-04 (Actual); Primary Completion 2020-09-30 (Actual); Study Completion 2020-09-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: James R McKay, PhD, Principal Investigator — University of Pennsylvania
Locations (3):
- United States (3):
  - Philadelphia VA Medical Center, Philadelphia, Pennsylvania
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - VA Pittsburgh Health System, Pittsburgh, Pennsylvania

RESULTS

PARTICIPANT FLOW:
Groups:
- Standard Care: In this arm, veterans receive the care that they would receive had they not enrolled in the research. No one will receive less than standard care.
  Brief Intervention
- Prevention Intervention: An adaptive monitoring intervention, delivered through text messages and brief telephone calls, that can provide extended prevention services for veterans engaging in risky alcohol use. After a veteran receives a BI for risky drinking, we will monitor alcohol use for 4 weeks. Veterans who reduce alcohol use to safe levels will be placed in a monitoring track, which consists of tailored text messages and brief monthly telephone contacts. Conversely, veterans who continue to use alcohol at hazardous levels will be placed in a track that provides tailored text messages and more frequent telephone calls. These calls provide further prevention/intervention services to help the veteran reduce alcohol use. These services address motivational issues and identify more effective ways to cope with stress and other factors that trigger unsafe alcohol use. Information on the veteran's progress is used to guide the content of subsequent text messages and prevention interventions.
  Prevention Intervention
  Brief Intervention
Period: Overall Study
Arm/Group | Standard Care | Prevention Intervention
Started | 50 | 58
Completed | 18 | 31
Not Completed | 32 | 27

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Standard Care | Prevention Intervention | Total
Number analyzed (Participants) | 50 | 58 | 108
Age, Continuous [Mean (Standard Deviation); unit: years] | 59.8 (10.3) | 58.5 (11.6) | 59.1 (11.03)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 4 | 8
  Male | 46 | 54 | 100
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 2 | 4
  Not Hispanic or Latino | 46 | 55 | 101
  Unknown or Not Reported | 2 | 1 | 3
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 29 | 30 | 59
  White | 19 | 22 | 41
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 2 | 5 | 7
Region of Enrollment [Number; unit: participants]
  United States | 50 | 58 | 108

OUTCOME MEASURES:

1. Primary Outcome: Rates of Risky Drinking, Week 13
Description: The primary outcome measure will be rates of the presence of any risky drinking in each week (i.e., more than 4 drinks per drinking day) as reported on the Time Line Follow Back.
Time Frame: weeks 1 - 13
Population: The analysis only includes participants for whom the data during this time period is complete. In addition, due to our finding that patients were unwilling to initially disclose alcohol use at screening, we enrolled people who were not necessarily drinking but monitored them. Once they began drinking they were received the intervention (or standard care) and were included in the analyses. However, many enrolled participants were not active drinkers and were not included in the analyses.
Measure: Mean (Standard Deviation); unit: risky drinking weeks
Arm/Group | Standard Care | Prevention Intervention
Number analyzed (Participants) | 15 | 44
risky drinking weeks | 3.03 (0.83) | 2.46 (0.65)

2. Primary Outcome: Rates of Risky Drinking, Week 26
Description: Rates of the presence of any risky drinking in each week (14 - 26)
Time Frame: weeks 14 - 26
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: risky drinking weeks
Arm/Group | Standard Care | Prevention Intervention
Number analyzed (Participants) | 15 | 38
risky drinking weeks | 2.97 (0.76) | 2.15 (0.55)

3. Primary Outcome: Rates of Risky Drinking, Week 39
Description: Rates of the presence of any risky drinking in each week (27 - 39)
Time Frame: weeks 27 - 39
Measure: Mean (Standard Deviation); unit: risky drinking weeks
Arm/Group | Standard Care | Prevention Intervention
Number analyzed (Participants) | 15 | 23
risky drinking weeks | 2.96 (0.79) | 2.44 (0.65)

4. Primary Outcome: Rates of Risky Drinking, Week 52
Description: Rates of the presence of any risky drinking in each week (40 - 52)
Time Frame: weeks 40 - 52
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: risky drinking weeks
Arm/Group | Standard Care | Prevention Intervention
Number analyzed (Participants) | 15 | 23
risky drinking weeks | 3.85 (1.03) | 2.50 (0.66)

5. Primary Outcome: Rates of Risky Drinking, Week 78
Description: Rates of the presence of any risky drinking in each week (53 - 78)
Time Frame: weeks 53 - 78
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: risky drinking weeks
Arm/Group | Standard Care | Prevention Intervention
Number analyzed (Participants) | 15 | 23
risky drinking weeks | 4.60 (1.31) | 2.70 (0.91)

ADVERSE EVENTS:
Time Frame: Adverse event data was collected for 18 months.
Arm/Group | Standard Care | Prevention Intervention
All-Cause Mortality (participants affected / at risk) | 3/50 | 0/58
Serious Adverse Events (participants affected / at risk) | 4/50 | 8/58
Other Adverse Events (participants affected / at risk) | 0/50 | 1/58
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Standard Care (N=50) | Prevention Intervention (N=58)
Hospitalized (Surgical and medical procedures) | 1 (2) | 4 (6)
hospitalized (Gastrointestinal disorders) | 1 (1) | 0 (0)
Hospitalized (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
hospitalized (General disorders) | 1 (1) | 0 (0)
ED visit (General disorders) | 1 (1) | 0 (0)
hospitalized (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
hospitalized (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Hospitalized (Cardiac disorders) | 0 (0) | 1 (2)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Standard Care (N=50) | Prevention Intervention (N=58)
emotional distress (Social circumstances) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-03-08): https://cdn.clinicaltrials.gov/large-docs/17/NCT02709317/Prot_SAP_000.pdf